CLINICAL TRIAL: NCT02240979
Title: Establishing a Non-invasive Method to Measure Heart Performance
Brief Title: Establishing a Non-invasive Method to Measure Your Heart's Performance
Status: Completed | Type: Observational
Sponsor: Marie Csete MD, PhD (Other)
Collaborators: University of Southern California (Other); California Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Marie Csete MD, PhD, Chief Scientific Officer, Huntington Medical Research Institutes
Organization: Huntington Medical Research Institutes (Other)
Other Study IDs: HMRI-10Pico-1; CIT2014 (Other: California Institute of Technology Boswell Fellowship)
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure
Keywords: arterial waveform; cardiac magnetic resonance imaging; echocardiography; intrinsic frequency measures of cardiac function
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults able to undergo cardiac MRI exam: Adults able to undergo cardiac MRI
  Interventions: Device: cardiac MRI

INTERVENTIONS:
Device: cardiac MRI — cardiac MRI

SUMMARY:
The purpose of the study is to evaluate a new way to examine cardiac function, using software developed at Caltech. The experimental device is software loaded on an iPhone. The iPhone is used to capture a pulse (waveform) by simply placing the iPhone lightly over the neck where the carotid pulse can be felt. In this study the information collected from the iPhone app is compared to cardiac function data obtained from the current gold standard for measuring cardiac function, cardiac magnetic resonance imaging (MRI). Subjects referred from cardiologists will also generally have echocardiography information available for comparison with the iPhone app. For the study, subjects will have completely non-invasive studies done in one setting: The iPhone app to capture the waveforms (over carotid and radial (wrist) arteries), tonometry (another non-invasive method using a modified stethoscope), standard pulse oximetry, followed by a 30 minute MRI examination of the heart. A second complete study will be done about 6 months after the first. The complete study session takes about 1.5 hours.

DETAILED DESCRIPTION:
Investigators at Caltech have developed an iPhone-based application that allows them to capture an arterial waveform using the iPhone camera held over the skin. Then based on the captured waveform and previous laboratory experiments and models, the investigators are able to calculate ejection fraction, the percentage of blood that goes out of the heart into the circulation with each beat. Previous studies suggested that the iPhone app measurements of ejection fraction were similar to those obtained with traditional cardiac echocardiography. In the current study the iPhone app measures are being compared to ejection fraction obtained using cardiac MRI. The iPhone also measures other physical properties of the heart and aorta that the investigators call "intrinsic frequencies". Using healthy subjects they have established the normal pattern/range of intrinsic frequencies, and in this study, a more diverse population of subjects (some with heart disease) will be studied, to determine how intrinsic frequency measures compare to traditional clinical measures of cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18-90, outpatients

Exclusion Criteria:

* Inability to lie flat for 30 minutes with periodic breath holding
* Metal implants or other standard contraindications to MRI
* Acute cardiac decompensation (active chest pain, shortness of breath)
* Hypotension (SBP<90 mm Hg)
* Claustrophobia
* Patient too large to fit in closed MRI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with normal and abnormal cardiac function will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance measures of cardiac function | Within 1 month of study
  Standard end-points of cardiac function such as chamber size and relaxation.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Csete, MD, PhD, Study Chair — Avicena LLC; Niema Pahlevan, PhD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Avicena LLC, Pasadena, California
  - Huntington Medical Research Institutes MR Imaging Center, Pasadena, California

IPD SHARING:
Plan to Share IPD: Yes
A manuscript was submitted in February 2016 reporting results of the study. In editorial process.

REFERENCES:
- [Background] Pahlevan NM, Tavallali P, Rinderknecht DG, Petrasek D, Matthews RV, Hou TY, Gharib M. Intrinsic frequency for a systems approach to haemodynamic waveform analysis with clinical applications. J R Soc Interface. 2014 Sep 6;11(98):20140617. doi: 10.1098/rsif.2014.0617. PMID 25008087
- [Derived] Niroumandi S, Rinderknecht D, Bilgi C, Cole S, Ogbonnaya SA, Wolfson AM, Vaidya AS, King KS, Pahlevan NM. Smartphone Measurement of Aortic Arch Pulse-Wave Velocity and Total Arterial Compliance: Accessible Local and Global Arterial Stiffness Assessment. J Am Heart Assoc. 2026 Feb 11:e043563. doi: 10.1161/JAHA.125.043563. Online ahead of print. PMID 41669977